CLINICAL TRIAL: NCT02820493
Title: Effectiveness of Vedolizumab Therapy in Inducing Clinical Remission in CD Patients Naïve to Anti-TNF and Its Capability to Halt Disease Progression
Brief Title: Effectiveness of Vedolizumab in CD Patients Naïve to Anti-TNF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Internal problems
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Giorgia Bodini, MD, PhD, Universita degli Studi di Genova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVeA Study
Record Dates: First submitted 2016-05-17; First posted 2016-07-01 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm study (Other): Vedolizumab 300 mg iv at week 0, week 2 and week 6, than every 8 weeks.
  Interventions: Drug: vedolizumab

INTERVENTIONS:
Drug: vedolizumab

SUMMARY:
Anti-cytokine antibodies, such as Infliximab (an anti TNF alfa chimeric antibody) and Adalimumab (an anti TNF alfa humanize antibody), have been developed and used in clinical practice for the treatment of patients with Crohn disease (CD). Unfortunately, their efficacy is limited. Based on these concepts, a new drug has been developed for IBD treatment. Vedolizumab (VDZ) is able to recognize the α4β7 heterodimer, and selectively blocks gut lymphocyte trafficking.

The hypothesis of this study is that VDZ therapy may be to halt CD disease progression during time and modifying its natural history, using Lemann Index.

DETAILED DESCRIPTION:
All patients who will enter in the study will be follow-up at weeks 2-6-14-22-30-38-46 or before in case of relapse. A relapse will be defined by an Harvey Bradshaw Index ≥ 5 for 2 consecutive weeks. The following data are to be recorded:

1. Physical examination
2. Adverse Event Review
3. Weight in Kg
4. Full blood count
5. Biochemical series including serum iron, serum ferritin, C reactive protein (PCR), ESR (eritrosedimatation rate)
6. Fecal Calprotectin
7. VDZ fecal loos
8. VDZ trough levels and antidrug antibodies
9. Current treatments

The last visit will be performed at week 54. The following data are to be recorded:

1. Physical examination
2. Adverse Event Review
3. Weight in Kg
4. Full blood count
5. Biochemical series including serum iron, serum ferritin, C reactive protein (PCR), ESR (eritrosedimatation rate)
6. Fecal Calprotectin
7. VDZ fecal loos
8. VDZ trough levels and antidrug antibodies
9. Current treatments
10. Routine lower and upper gastrointestinal endoscopy and magnetic resonance imaging or computed tomography of the small bowel
11. SES-CD
12. Lemann Index

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged between 18 and 80
* Have a moderate/severe CD defined by an HBI >7 CD

Exclusion Criteria:

* previous treatment with anti-TNF drugs,
* concomitant use of immune-modulator drugs for CD (azathioprine/6-mercaptopurine, methotrexate)
* ulcerative colitis (UC) or inflammatory bowel disease undetermined (IBD-U) diagnosis
* symptomatic obstructive disease
* bowel resection within the past 6 months
* ileostomy
* extensive small bowel resection (as determined by the investigator) or a short bowel syndrome
* patients who are currently receiving total parenteral nutrition
* history of cancer in the past 5 years
* pregnancy known at the study inclusion
* positive Clostridium difficile stool assay
* Listeria, human immunodeficiency virus, central nervous system demyelinating disease, untreated tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Harvey Bradshaw index | Week 0-14
  Primary responders will defined as by a decrease of Harvey Bradshaw Index at week 14 of 3 point from the Harvey Bradshaw Index calculate at week 0.

SECONDARY OUTCOMES:
Lèmann Index | Week 0 and Week 54
VDZ trough levels | Week 0-2-6-14-22-30-38-46-54
anti-drug antibodies | Week 0-2-6-14-22-30-38-46-54
fecal VDZ loss | Week 0-2-6-14-22-30-38-46-54
  The investigators will evaluated the VDZ quantity (microgram) that a patients with mucosal ulcers could loss in patients feces.